CLINICAL TRIAL: NCT05350254
Title: C-prior: Implementation of the MAINTAIN Instrument for Patients With Dysfunctional Spinal Pain - a Randomized Clinical Trial
Brief Title: Implementation of the MAINTAIN Instrument for Patients With Dysfunctional Spinal Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: Parker University (Other); Karolinska Institutet (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 222006
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Low Back Pain, Recurrent; Neck Pain; Back Pain
MeSH Terms: conditions — Low Back Pain; Neck Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stratified Maintenance Care (Experimental): All participating patients will receive pragmatic chiropractic care for the initial 3 weeks (6 visits) and home exercise recommendations.
  Participants in the Stratified Maintenance Care group will be classified based on the MAINTAIN instrument into: not a candidate, good candidate, and very good candidate for maintenance care:
  * Participants showing a good response to the initial care and classified as not a candidate or a good candidate for maintenance care will be given home exercise recommendations. Return for further manual treatment will be recommended if they have a relapse or exacerbation of symptoms (symptom-guided care).
  * Participants classified as having a good response to the initial care and very good candidates for maintenance care, will have visits with tapering manual treatments and home exercise recommendations. They will then be recommended maintenance care with pre-planned visits at 4-12 week intervals (aiming at increasing the interval as soon as possible).
  Interventions: Other: Chiropractic maintenance care
- Standard Chiropractic Care (Active Comparator): All participating patients will receive pragmatic chiropractic care for the initial 3 weeks (6 visits) and home exercise recommendations.
  In the Standard chiropractic care group, participating patients will receive a standard (pragmatic) chiropractic care in which treatment will be provided based on the clinician's judgement and home exercise recommendations. This may or may not include maintenance care depending on the clinicians' standard operating procedures. All treatments provided will be recorded. Return for further treatment will be recommended if they have a relapse or exacerbation of symptoms (symptom-based).
  Interventions: Other: Standard chiropractic care

INTERVENTIONS:
Other: Chiropractic maintenance care — Manual Therapy, individual exercises and lifestyle advice
  Arms: Stratified Maintenance Care
Other: Standard chiropractic care — Standard care based on clinician's judgement
  Arms: Standard Chiropractic Care

SUMMARY:
Previous studies showed that some back pain patients (with specific characteristics) present less days with pain when treated with chiropractic maintenance care. A clinical instrument (called MAINTAIN instrument) was developed to identify those patients who would benefit from chiropractic maintenance care. This study will investigate the impact of using the MAINTAIN instrument in clinical practice. This study will help to improve clinical care of patients with back and neck pain by providing them with more individualized care.

DETAILED DESCRIPTION:
Rationale: Non-specific Low Back Pain (LBP) is one of the largest societal economic burdens with a 80-85% lifetime prevalence worldwide, often characterized by recurrent episodes. Chiropractic maintenance care (MC) is a management strategy aimed at preventing LBP episodes and deterioration by treating patients at pre-planned intervals, regardless of symptoms. It consists of manual therapy, individual exercises and lifestyle advice, and patients are selected based on their previous history of pain and the effectiveness of the initial care plan. A pragmatic randomized clinical trial showed that patients receiving MC had 12.8 fewer days with bothersome LBP compared to a control group. More specifically, patients in the Dysfunctional sub-group, categorized by the West Haven-Yale Multidimensional Pain Inventory (MPI) instrument, reported fewer days with pain when receiving MC, suggesting MC's superior effectiveness in this subgroup of patients. The MPI instrument, however, is not suited for daily clinical practice use, prompting the development of the more practical MAINTAIN instrument. It captures 5 dimensions of the pain experience yielding 3 categories of patients: not a candidate for MC, good candidate for MC (sensitivity: 95.8%; specificity: 64.3%) and very good candidate for MC (sensitivity: 81.1%; specificity: 79.2%). Despite these encouraging preliminary results, the usability and impact of using the MAINTAIN instrument in clinical practice remains unknown and a thorough investigation on its implementation is fundamental.

Purpose: The overall goal of this multicenter randomized clinical trial is to investigate the process and outcomes of implementing the MAINTAIN instrument in clinical practice. The specific aims are to: 1) assess the effectiveness and cost-effectiveness of stratified MC using the MAINTAIN instrument compared to standard chiropractic care; and 2) assess the fidelity and procedure compliance of implementing the MAINTAIN instrument.

Analysis Plan: An intention to treat protocol will be used and estimates will be reported with arithmetic means and 95% confidence intervals. Analysis of the primary outcome (number of days with activity limiting pain) will be conducted as it was in Eklund et al. (2018, 2019). The total number of days with activity limiting pain will be modelled using Generalized Estimating Equations (GEE) linear regression, using appropriate correlation structure and robust variance estimator. Terms for study arm, time and study arm by time interaction will be included. A term for MC candidate (Yes or No) will be added to this model to further investigate the stratification and its relationship to outcomes. The RE-AIM framework will be used to assess the impact and implementation of the MAINTAIN instrument.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spinal pain (neck, mid-back, and/or low back) of recurrent (not the first episode) and significant (more than 30 days in the past 12 months) character
* No pain episode in the past 3 months
* Access to a mobile phone and email.
* Ability to send and receive SMS (text messages).

Exclusion Criteria:

* Pregnancy
* Serious pathology (e.g., acute trauma, cancer, infection, cauda equina, osteoporosis, vertebral fractures)
* Contraindications to manual therapy
* Specific spinal conditions (e.g., radiculopathy, spinal stenosis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of days with activity-limiting pain | 12-months
  Number of days with activity-limiting pain

SECONDARY OUTCOMES:
Number of missed working days | 12-months
  Number of missed working days due to pain
Loss of work productivity | 12-months
  11-point numeric rating scale, where 0 = did not affect my work and 10 = completely prevented me from working
Pain intensity | 12-months
  11-point visual analogue scale, where 0 = no pain and 100 = worst imaginable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Canadian Memorial Chiropractic College, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This study will be part of an international project where multiple coordinated trials will collect data on different aspects of maintenance care. While this specific project is independent and focuses on Canadian population, a core set of outcomes collected in each study will be merged with data from the other trials internationally for secondary analyses.

REFERENCES:
- [Derived] Funabashi M, Ives G, Pohlman KA, Hogg-Johnson S, Townsend M, Macedo L, Lee J, Eklund A. C-prior-implementation of the MAINTAIN instrument for patients with spinal pain: study protocol for a randomized clinical trial. Trials. 2026 Feb 10. doi: 10.1186/s13063-026-09509-6. Online ahead of print. PMID 41664083